CLINICAL TRIAL: NCT01431729
Title: Honey and a Mixture of Honey, Beeswax and Olive Oil-propolis Extract in Treatment of Chemotherapy-induced Oral Mucositis: a Randomized Controlled Pilot Study
Brief Title: Honey and a Mixture of Honey, Beeswax and Olive Oil-propolis Extract in Treatment of Chemotherapy-induced Oral Mucositis
Status: Completed | Type: Observational
Sponsor: mamdouh abdulmaksoud abdulrhman (Other)
Responsible Party: Sponsor-Investigator, mamdouh abdulmaksoud abdulrhman, professor of pediatrics, faculty of medicine, ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: honey propolis 421
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Honey

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- mucositis
  Interventions: Other: honey, hope,mucositis

INTERVENTIONS:
Other: honey, hope,mucositis — Eligible patients were randomly allocated by a computer-generated list of random numbers to be assigned into one of three treatment groups; Group (1) received an empirical dose of 15 gm honey applied topically to the affected oral mucosa three times daily until healing or for 10 days, which ever comes first. Group (2) received an empirical dose of 5 gm of a 4:2:1 mixture of honey, olive oil-propolis extract and beeswax (HOPE) applied topically to the oral mucosa three times daily until healing or for 10 days, which ever comes first. Group (3) served as controls and received benzocaine 7.5% gel applied topically to areas of ulcers three times daily.
  Other Names: honey,propolis,olive oil, mucositis

SUMMARY:
Although, oral mucositis has been studied for many years, no available treatment has been shown to be effective in preventing or treating mucositis. Based on the observations that honey and other products of honeybees have anti-inflammatory, anti-oxidant, anti-microbial and wound healing effects, the present study aims at evaluation of the effect of topical application of honey and a mixture of honey, beeswax and olive oil-propolis extract, as natural products, in treatment of chemotherapy-induced oral mucositis in children with acute lymphoblastic leukemia (ALL). This is a randomised controlled clinical trial in which eligible patients were randomly assigned into three equal treatment groups. Group 1 received 15 gm honey applied topically to the affected oral mucosa three times daily. Group 2 received 5 gm of a mixture of honey, olive oil-propolis extract and bees wax (HOPE) applied topically to the oral mucosa three times daily. Group 3 served as control and received a 7.5% benzocaine gel applied to the areas of ulcers three times daily.

DETAILED DESCRIPTION:
All patients with ALL during the consolidation phase of treatment, and with chemotherapy-related oral mucositis grades 2 and 3 were candidates for this trial.Exclusion criteria included the presence of any of the following: (1) coexisting diabetes mellitus, (2) administration of antiviral, antifungal therapy and / or any other treatment for oral mucositis before enrollment in the study, (3) presence of neutropenia (absolute neutrophilic count [ANC] ≤ 1500/mm3), (4) presence of advanced or severe periodontitis (patients with periodontal pockets of 6 mm or more. The primary outcome measure was the "recovery time", defined as the number of days from initiation of treatment to when complete healing of all ulcers occurred.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ALL during the consolidation phase of treatment, and
* with chemotherapy-related oral mucositis grades 2 and 3

Exclusion Criteria:

1. coexisting diabetes mellitus,
2. administration of antiviral, antifungal therapy and / or any other treatment for oral mucositis before enrollment in the study,
3. presence of neutropenia (absolute neutrophilic count [ANC] ≤ 1500/mm3),
4. presence of advanced or severe periodontitis (patients with periodontal pockets of 6 mm or more)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients were randomly allocated by a computer-generated list of random numbers to be assigned into one of three treatment groups; 30 patients each. Group (1) received an empirical dose of 15 gm honey applied topically to the affected oral mucosa three times daily until healing or for 10 days, which ever comes first. Group (2) received an empirical dose of 5 gm of a 4:2:1 mixture of honey, olive oil-propolis extract and beeswax (HOPE) applied topically to the oral mucosa three times daily until healing or for 10 days, which ever comes first. Group (3) served as controls and received benzocaine 7.5% gel applied topically to areas of ulcers three times daily.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
"Recovery time" , defined as the number of days from initiation of treatment to when complete healing of all ulcers will occur. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh Abdulrhman, professor, Principal Investigator — professor
Locations (1):
- Hematology - Oncology, Children's Hospital, Ain Shams University, Cairo, Abbasia, Egypt

REFERENCES:
- [Derived] Abdulrhman M, Elbarbary NS, Ahmed Amin D, Saeid Ebrahim R. Honey and a mixture of honey, beeswax, and olive oil-propolis extract in treatment of chemotherapy-induced oral mucositis: a randomized controlled pilot study. Pediatr Hematol Oncol. 2012 Apr;29(3):285-92. doi: 10.3109/08880018.2012.669026. PMID 22475306
- See also: mamdouh565@hotmail.com — http://www.shams.edu.eg/